CLINICAL TRIAL: NCT04707677
Title: Comparative Aesthetic Analysis Between Titanium and Ceramic Implants: A 12-month Randomized Clinical Trial.
Brief Title: Comparative Aesthetic Analysis Between Titanium and Ceramic Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Santiago de Compostela (Other)
Responsible Party: Principal Investigator, Juan Blanco Carrión, Doctorate in Dentistry, University of Santiago de Compostela
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CI_RCT_US16
Record Dates: First submitted 2021-01-10; First posted 2021-01-13 (Actual); Last update posted 2021-12-27 (Actual); Status verified 2021-02

CONDITIONS: Dental Implants

STUDY DESIGN:
Intervention Model Description: Two study groups, test (titanium implants) and control (ceramic implants)
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CONTROL GROUP (Active Comparator): Implant surgery placement. Tissue Level SLA Titanium implant (Straumann Standard Plus Narrow Neck CrossFit®; Institut Straumann, Basel, Switzerland). The implant had a diameter of 3.3 mm and a polished neck of 1.8 mm. The length of the implants was 8, 10 and 12 mm and was chosen according to the patient's anatomy.
  Interventions: Device: Titanium and ceramic dental Implants
- TEST GROUP (Experimental): Implant surgery placement. Tissue Level Ceramic monotype implant was placed (Straumann PURE Ceramic implants®; Institut Straumann, Basel, Switzerland). The implant had a diameter of 3.3 mm and a polished neck of 1.8 mm. The length of the implants was 8, 10 and 12 mm and was chosen according to the patient's anatomy.
  Interventions: Device: Titanium and ceramic dental Implants

INTERVENTIONS:
Device: Titanium and ceramic dental Implants — Two types of implant placement and follow-up to compare the esthetic, clinical and radiographic parameters between them.

SUMMARY:
Objective: The aim of this randomized clinical trial was to compare ceramic and titanium implants with respect to the esthetic and clinical parameters, and patient reported outcome measures (PROMs).

Material and methods: Thirty patients received thirty implants (8-12 mm in length, 3.3 mm diameter and a tissue level design) to replace the absence of a single tooth in the anterior maxilla. Patients were randomly allocated to receive a ceramic or a titanium implant. Esthetic and clinical parameters and PROMs were evaluated 18 months after surgery.

DETAILED DESCRIPTION:
The study was a double-blind randomized controlled clinical trial (RCT), with a parallel design, comparing ceramic (test group) and titanium (control group) implants, for the replacement of a single-tooth in the anterior maxilla.

All patients were randomized and assigned to each of the study groups through a computer-generated randomization.

Surgical and restorative procedures In the test group, a Tissue Level Ceramic monotype implant was placed (Straumann PURE Ceramic implants®; Institut Straumann, Basel, Switzerland) and in the control group a Tissue Level SLA Titanium implant (Straumann Standard Plus Narrow Neck CrossFit®; Institut Straumann, Basel, Switzerland). The length of the implants was 8, 10 and 12 mm.

The primary outcome was the Implant Crown Aesthetic Index (ICAI). It consists of nine sections: mesiodistal dimension of the crown, position of the incisal edge of the crown, labial convexity of the crown, color and translucency of the crown, crown surface, position of the gingival margin of the peri-implant mucosa, position of the interdental papilla, contour of the vestibular mucosa and color and surface of the vestibular mucosa. These sections were compared with the adjacent and contralateral tooth as a reference and assigned the following score: 0, excellent; 1 or 2 satisfactory; 3 or 4 moderate; 5 or more bad.

ELIGIBILITY:
Inclusion Criteria:

* Periodontal and systemically healthy patients > 18 years of age, with good plaque control (< 25%).
* Patients with a missing tooth in the anterior maxilla (from 13 to 23) with the presence of adjacent natural dentition mesially and distally (single gap). A minimum of 4 months of healing after tooth extraction was required before implant insertion.
* Presence of ≥ 2mm of keratinized tissue.
* Simultaneous bone regeneration was allowed during surgery.

Exclusion Criteria:

* Intake any medication or presence of any systemic disease that could affect bone metabolism.
* Pregnancy, or lactating women.
* Active periodontal disease
* Smoking >10 cig/day

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-09-15 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
The primary outcome was the Implant Crown Aesthetic Index (ICAI). | 36 months
  It consists of nine sections: (i) mesiodistal dimension of the crown, (ii) position of the incisal edge of the crown, (iii) labial convexity of the crown, (iv) color and translucency of the crown, (v) crown surface, (vi) position of the gingival margin of the peri-implant mucosa, (vii) position of the interdental papilla, (viii) contour of the vestibular mucosa and (ix) color and surface of the vestibular mucosa. These sections were compared with the adjacent and contralateral tooth as a reference and assigned the following score: 0, excellent; 1 or 2 satisfactory; 3 or 4 moderate; 5 or more bad (Meijer et al., 2005).

CONTACTS AND LOCATIONS:
Overall Officials: Juan Blanco, Study Director — University of Santiago de Compostela
Locations (1):
- Master Periodoncia, Santiago de Compostela, Spain

IPD SHARING:
Plan to Share IPD: No